CLINICAL TRIAL: NCT01660386
Title: An Open-label, Randomized, Four-way Cross-over, Single Dose Study to Compare the Different Effect of DPP-4 Inhibitors and Sulfonylurea on the Beta Cell Function by Using "Biphase-Hyperglycemic Clamp"
Brief Title: Study of Comparing the Different Effect of DPP-4 Inhibitors and Sulfonylurea by Using "Biphase-Hyperglycemic Clamp"
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, the vice-president of Shanghai Jiao Tong University affiliated Rui jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CCEMD014
Record Dates: First submitted 2012-08-05; First posted 2012-08-08 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Dpp-4 inhibitor; Sulfonylurea; beta cell function
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; saxagliptin; glimepiride; BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sitagliptin (Experimental): the subjects are asked to take one pill of sitagliptin(100mg po once) in 7am of experimental day then start bi-phase hyperglycaemic clamp at 9am.
  Interventions: Drug: Sitagliptin
- Saxagliptin (Experimental): the subjects are asked to take one pill of saxagliptin(5mg po once) in 7am of experimental day then start bi-phase hyperglycaemic clamp at 9am.
  Interventions: Drug: Saxagliptin
- Glimepiride (Experimental): the subjects are asked to take one pill of glimepiride(2mg po once) in 7am of experimental day then start bi-phase hyperglycaemic clamp at 9am.
  Interventions: Drug: Glimepiride
- Blank control (Other): the subjects take no medication at experimental day and start bi-phase hyperglycaemic clamp at 9am.
  Interventions: Drug: Blank control

INTERVENTIONS:
Drug: Sitagliptin — 100mg po once
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Saxagliptin — 5mg po once
  Other Names: Onglyza
  Arms: Saxagliptin
Drug: Glimepiride — 2mg po once
  Other Names: Amaryl
  Arms: Glimepiride
Drug: Blank control — the subjects take no medication at experimental day and start bi-phase hyperglycaemic clamp at 9am.
  Other Names: Baseline
  Arms: Blank control

SUMMARY:
The objective of this study is to demonstrate the different effects of two DPP-4 inhibitors(Sitagliptin, Saxagliptin)and the insulin secretagogue: glimepiride on first and second phase insulin secretion by using a Biphase-Hyperglycemic Clamp and to explore the different effects of the study drugs on the GLP-1 response, and the glucagon concentration which indicates alpha cell function in healthy subjects.

DETAILED DESCRIPTION:
After enrollment and two weeks screening period eligible subjects will be counseled to follow a dietary program for approximately 2 wk and recorded of personal history, full clinical examination and screening blood samples.

Subjects will be randomized using a computer-generated allocation schedule to one of 12 sequences during which each subjects will be assigned to take 4 times of bi-phase hyperglycaemic clamp experiments at a randomized sequence separated by a washout period of 7-14d.

At each experimental day, the subject will take the given dose of Sitagliptin, Saxagliptin, Glimepiride and nothing for blank control two hours before the clamp experiment starts.

The hyperglycaemic clamp will be performed after an overnight fast. Subjects will be placed in a recumbent position and cannula will be inserted in a dorsal hand vein. The hand will be placed in a heating box (42C) throughout the experiment to allow frequent sampling of arterialized blood. A second cannula will be inserted in a contralateral cubital vein for glucose infusion.

At time zero (0 min), a 50% glucose bolus will be injected during 1 min to increase PG to 12mM. The glucose bolus will be calculated as:(12mM-FPG)×35 mg glucose × body weight (kg). PG will be measured bedside every 5 min and maintained at 12mM by an adjustable continuous 20% glucose infusion. After 90min, PG will be lowered down below 6mM for the islet cells to rest, then the subject will be instructed to consume 75g glucose solution orally in 5min, PG will be measured bedside every 5 min and maintained below 6mM for 40min then restart the 90min-hyperglycaemic clamp experiment. The oral period of hyperglycaemic clamp process is the same as what's done in fasting period. Blood samples will be collected in -2h, 0min, 10min, 90min in both hyperglycaemic clamp experimental process for the measurement of insulin, C-peptide, glucagon, active GLP-1, total GLP-1 and DPP-4 activity.

Thus we could evaluate the beta cell function represented by the first phase and the second phase of insulin secretion(C-peptide secretion) and alpha cell function represented by the change of glucagon concentration during the fasting period and oral period of hyperglycaemic clamp experiment and the change of active GLP-1, total GLP-1 and DPP-4 activity as well.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted;
2. Having good study compliance;
3. Healthy Male subjects between 20-30 years of age (inclusive), and in good health as determined by past medical history, physical examination, vital signs, and clinical laboratory test;
4. Must have a body mass index (BMI) between 19-25kg/m2 (inclusive);
5. No weight fluctuation greater than 5% in late 3 months。

Exclusion Criteria:

1. With impaired glucose tolerance, T2DM or any significant medical condition (within 3 years), laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study;
2. Used any prescribed systemic or topical medication within 30 days of the first dose administration;
3. Any medical or surgical conditions possibly affecting study drug absorption, distribution, metabolism and excretion;
4. Participated in a clinical study involving administration of an investigational drug within 90 days preceding the first dose administration or within five half-lives of the first dose administration (whichever is longer);
5. Donated blood or plasma or had any other significant blood loss within 2 months preceding the first dose administration;
6. History of multiple drug allergies;
7. Any clinically significant allergic disease;
8. Recently drug or alcohol abuse (>35 unit/week, 1 unit=8g alcohol @ 1 standard drink @ 250ml beer @ 140ml wine @ 25ml strong alcohol drink like whiskey);
9. Smokers or users of other tobacco products in the 3 months prior to screening.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
The acute phase and second phase of insulin secretion and C peptide secretion | 1-2 months
  The primary outcome measures are improvement in beta cell function measured as insulin secretion and C-peptide secretion during the bi-phase hyperglycaemic clamp. The first phase of insulin and C-peptide secretion is defined as the secretion between 0-10min, the second phase is defined as secretion between 20-90min of bi-phase hyperglycaemic clamp

SECONDARY OUTCOMES:
Alpha cell function,GLP-1 response | 1-2 months
  The secondary outcome measures are a relative increase in glucagon concentration which indicates alpha cell function and the GLP-1 response, DPP-4 activity and before taken the medicine and in 0, 10, 90,150,160,240min during the bi-phase hyperglycaemic clamp.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD. PHD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Shanghai, China